CLINICAL TRIAL: NCT03186638
Title: Phase II Study of Low-Dose Ibuprofen for Cognitive Problems in Patients With Cancer
Brief Title: Low-Dose Ibuprofen in Improving Cognitive Impairment in Patients With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michelle Janelsins, PhD, MPH, Associate Professor, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: URCC16092; NCI-2017-00790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC16092 (Other: University of Rochester NCORP Research Base); URCC-16092 (Other: DCP); URCC-16092 (Other: CTEP); R21CA187500 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Impairment; Malignant Neoplasm
MeSH Terms: conditions — Cognitive Dysfunction; Neoplasms | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ibuprofen) (Experimental): Patients receive ibuprofen PO BID for 6 weeks.
  Interventions: Drug: Ibuprofen; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 6 weeks.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Ibuprofen — Given PO
  Other Names: (.+ -.)-p-Isobutylhydratropic acid; Advil; Motrin; p-Isobutylhydratropic acid
  Arms: Arm I (ibuprofen)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well low-dose ibuprofen in improving cognitive impairment in patients with cancer. Anti-inflammatory agents, such as ibuprofen, may slow the decline of cognitive processes and diseases involving the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide preliminary data on the effect of ibuprofen on alleviating chemotherapy-related cognitive impairment (CRCI) in cancer patients receiving chemotherapy or who have received chemotherapy within the last 6 months compared to a placebo control, as assessed by the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog).

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients receive ibuprofen orally (PO) twice daily (BID) for 6 weeks.

ARM II: Patients receive placebo PO BID for 6 weeks.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer and have had surgery and are now receiving adjuvant or neoadjuvant chemotherapy or who have received chemotherapy within the last 6 months; chemotherapy with concurrent radiation therapy (RT) is allowed
* Answer YES to the question: "Have you noticed any problems in your memory, attention, concentration, multi-tasking or other cognitive functions?" any time after initiation of chemotherapy cycle 1

  * NOTE: If a participant answers NO, they may be re-approached at a subsequent cycle
* Be able to swallow medication
* Be able to read English
* Have the ability to understand and to give written informed consent as assessed by the participant's primary care physician or medical oncologist

Exclusion Criteria:

* Have a confirmed brain tumor or brain metastases
* Be taking a regular daily dose of an NSAID NOTE: Daily doses of 81 mg aspirin are permitted and higher doses of an NSAID on an 'as needed' basis are permitted
* Be diagnosed with dementia or severe neurodegenerative disease
* Have a contraindication to NSAIDs at the oncologist's discretion (i.e., allergy, worsening of ongoing medical problem due to NSAID, very low platelet count from chemotherapy, full-dose anti-coagulation/high risk of bleeding, and uncontrolled conditions such as hypertension, asthma, or peptic ulcer disease)
* Have been hospitalized for treatment of a major psychiatric illness within the last five years
* Have a serum creatinine above 1.5 upper limit of normal (ULN) (collected within the past 4 weeks); ULN is per institutional definition
* Concurrent administration of warfarin, full dose aspirin, clopidogrel, apixaban or other medications known to increase the risk of bleeding or to interfere with antiplatelet activities
* Be colorblind
* Have active substance abuse (e.g. alcohol, drugs) per self-report or medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Janelsins, Principal Investigator — University of Rochester NCORP Research Base
Locations (169):
- United States (169):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Bronson Battle Creek, Battle Creek, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Marietta Memorial Hospital, Columbus, Ohio
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Greenville Health System Cancer Institute-Laurens, Clinton, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Ibuprofen) | Arm II (Placebo)
Started (Randomized) | 45 | 42
Received Intervention and Completed Baseline Assessments | 44 | 40
Completed | 37 | 36
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Withdrawn due to medical problem | 3 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ibuprofen 200mg BID: 200mg ibuprofen (taken twice a day at least 8 hours apart) for a period of 6 weeks.
  Ibuprofen: 200 mg BID and 8 hours apart
- Placebo: 200mg placebo (taken twice a day at least 8 hours apart) for a period of 6 weeks.
  Placebo: 200mg BID and 8 hours apart
- Total: Total of all reporting groups
Arm/Group | Ibuprofen 200mg BID | Placebo | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (12.5) | 54.6 (12.8) | 55 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 41 | 38 | 79
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 40 | 37 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Cancer Type [Count of Participants; unit: Participants]
  Breast | 20 | 20 | 40
  Colorectal | 14 | 11 | 25
  Other | 10 | 11 | 21
  Unknown or Not Reported | 1 | 0 | 1
Education Level [Count of Participants; unit: Participants]
  Some High School or Less | 1 | 0 | 1
  Highschool/GED | 9 | 5 | 14
  Less than 4 Year Degree | 9 | 11 | 20
  4 Year Degree | 16 | 12 | 28
  Graduate Degree | 9 | 12 | 21
  Unknown or Not Reported | 1 | 2 | 3
Cancer Stage [Count of Participants; unit: Participants] — Stage 1.This stage is usually a small cancer or tumor that has not grown deeply into nearby tissues. It also has not spread to the lymph nodes or other parts of the body.
  Stage 2 and 3.These stages indicate larger cancers or tumors that have grown more deeply into nearby tissue. They may have also spread to lymph nodes but not other parts of the body.
  Stage 4.This stage means that the cancer has spread to other organs or parts of the body. It may also be called metastatic cancer.
  Stage 1 is best, Stage 4 is worst.
  Participants
    Stage 1 | 7 | 2 | 9
    Stage 2 | 8 | 13 | 21
    Stage 3 | 16 | 12 | 28
    Stage 4 | 10 | 11 | 21
    Unknown or Not Reported | 4 | 4 | 8
Chemotherapy [Count of Participants; unit: Participants]
  Actively Receiving | 37 | 34 | 71
  Not Actively Receiving | 7 | 8 | 15
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Effects of Ibuprofen on Alleviating Chemotherapy-related Cognitive Impairment
Description: Will be assessed by the Functional Assessment of Cancer Therapy-Cognitive Function. Means, standard deviations, and 95% confidence intervals will be determined in order to estimate preliminary population variances and effect sizes. These statistical measures will be calculated by group for the Pre(Baseline) and Post(6 Weeks) measures of the Functional Assessment of Cancer Therapy-Cognitive Function scores as well as the change (post-pre) in the scores using the subjects that completed the study (complete case estimation). The complete case estimates will be compared to multiple imputation estimates based on all subjects that completed pre-intervention. An analysis of covariance will be run using Functional Assessment of Cancer Therapy-Cognitive Function post-intervention as the response. Higher scores indicate better function; range is 0 to 148.
Time Frame: Up to 41 days post-intervention
Population: Whenever the 6-week number of subjects or baseline number of subjects is less than the number reported per arm this is due to the data not being available. n=36 for Placebo (3-withdrawal by subject, 1- withdrawal due to medical issue) ; n=37 for Ibuprofen (3-withdrawal by subject, 3 - withdrawal due to medical issue, 1-lost to follow-up*)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ibuprofen 200 mg BID: 200mg ibuprofen (taken twice a day at least 8 hours apart) for a period of 6 weeks.
  Ibuprofen: 200 mg BID and 8 hours apart
Arm/Group | Ibuprofen 200 mg BID | Placebo
Number analyzed (Participants) | 44 | 40
score on a scale
  Baseline (Pre) | 89.98 (27.82) | 91.08 (25.98)
  6 Weeks (Post): number analyzed (Participants) | 37 | 36
  6 Weeks (Post) | 105.54 (25.44) | 107.75 (24.83)
  Change from Baseline(Post - Pre): number analyzed (Participants) | 37 | 36
  Change from Baseline(Post - Pre) | 14.59 (22.02) | 15.52 (21.43)
Statistical Analysis 1: Comparison: Ibuprofen 200 mg BID vs Placebo; Test type: Superiority; p = 0.7917, ANCOVA; Adjusted for Baseline values

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study intervention period. Approximately 6 weeks
Description: Adverse event definition does not differ from clinicaltrials.gov definition. A serious adverse event (SAE) is any adverse event, occurring at any dose and regardless of causality that: Results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, or is an important medical event.
Arm/Group | Ibuprofen 200 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/42
Serious Adverse Events (participants affected / at risk) | 2/45 | 3/42
Other Adverse Events (participants affected / at risk) | 15/45 | 15/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen 200 mg BID (N=45) | Placebo (N=42)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen 200 mg BID (N=45) | Placebo (N=42)
Anemia (Blood and lymphatic system disorders) | 3 (7) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Chest wall pain (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Anemia (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0)
Thromboembolic Event (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT03186638/Prot_SAP_000.pdf